CLINICAL TRIAL: NCT04874259
Title: Effectiveness of Liver Transplantation for Unresectable Colorectal Liver Metastasis; Pilot Study
Brief Title: LT for Unresectable Colorectal Liver Metastasis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Nam-Joon Yi, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 209-176-1162
Record Dates: First submitted 2021-05-02; First posted 2021-05-05 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Liver Metastasis Colon Cancer
Keywords: colorectal cancer; liver metastasis; living donor liver transplantation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Colorectal cancer liver metastasis (Experimental): Liver transplantation for the treatment of unresectable colorectal cancer liver metastasis
  Interventions: Procedure: Living donor liver transplantation

INTERVENTIONS:
Procedure: Living donor liver transplantation — Living donor liver transplantation

SUMMARY:
Unlike hepatocellular carcinoma, liver transplantation in patients with liver metastasis from colorectal cancer is limited in only few centers. Previously, it was not generally implemented due to lack of organs and high recurrence rates after transplantation. However, due to progressive development in treatments, good results such as increased survival rates can be expected even in liver transplant patients with liver metastasis from colorectal cancer, which is known to have poor prognosis. Therefore, the purpose of this study is to analyze the efficacy of liver transplantation as an alternative treatment for liver metastasis from colorectal cancer.

DETAILED DESCRIPTION:
Surgical treatment offers a distinct survival benefit in liver metastasis of colorectal cancer (CRC LM). However, it has been estimated that only 40% of patients are candidates for curative liver resection. Liver transplantation can be considered as one of a treatment option, since all evident disease is removed during procedure. However, it is limited in only few centers due to lack of organs and high recurrence rates after transplantation.

Currently, with help of development in treatments, prognosis after LT in CRC LM is improving. Recent study of LT for CRC LM from Norway demonstrated a 5-year survival of 56%. In addition, cohort study and randomized controlled trials are ongoing in Germany and Canada. Therefore, it seems to be necessary to verify the effectiveness of liver transplantation for CRC LM and to verify it as an alternative treatment if there is no other treatment. The purpose of this study is to analyze the efficacy of liver transplantation as an alternative treatment for liver metastasis from colorectal cancer.

Potential participants will be evaluated for liver transplantation and must also have a willing, healthy living donor. Unresectable metastasis should be limited to the liver and stable without no other treatment such as immunotherapy, chemotherapy, surgical resection, and radiofrequency ablation. The suitability of liver transplantation will be evaluated through a multidisciplinary assessment immediately before transplantation. Those participants who undergo liver transplantation will be followed for survival, disease-free survival, and recurrence for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Proven colorectal cancer liver metastases without no other treatment (such as immunotherapy, chemotherapy, surgical resection, and radiofrequency ablation)
* Metastasis isolated to liver
* Patients selected as a liver transplant recipient at a multidisciplinary meeting
* Paitents with a willing, healthy living donor
* Willing and able to provide written informed consent

Exclusion Criteria:

* Pregnant women
* Known history of human immunodeficiency virus (HIV) infection
* Patients with active peptic ulcer within 2 weeks of transplantation
* Persistent colorectal cancer after colon resection
* Hemodynamically unstable prior to liver transplantation
* Progression of LM at any timepoint prior to transplant surgery (assessed in a multidisciplinary meeting)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
1 year patient survival | 1 year
  1 year patient survival

SECONDARY OUTCOMES:
1 year disease-free survival | 1 year
  1 year disease-free survival
3 year patient survival | 3 year
  3 year patient survival
3 year disease-free survival | 3 year
  3 year disease-free survival
Recurrence | 3 year
  Site and pattern of recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Nam-Joon Yi, Ph.D., Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koffron A, Fryer JP, Abecassis M. Indications and results of liver transplantation for primary and metastatic liver cancer. Cancer Treat Res. 2001;109:77-99. doi: 10.1007/978-1-4757-3371-6_5. No abstract available. PMID 11775446
- [Background] Honore C, Detry O, De Roover A, Meurisse M, Honore P. Liver transplantation for metastatic colon adenocarcinoma: report of a case with 10 years of follow-up without recurrence. Transpl Int. 2003 Sep;16(9):692-3. doi: 10.1007/s00147-003-0605-3. Epub 2003 Jun 12. PMID 12802483
- [Background] Kappel S, Kandioler D, Steininger R, Langle F, Wrba F, Ploder M, Berlakovich G, Soliman T, Hetz H, Rockenschaub S, Roth E, Muhlbacher F. Genetic detection of lymph node micrometastases: a selection criterion for liver transplantation in patients with liver metastases after colorectal cancer. Transplantation. 2006 Jan 15;81(1):64-70. doi: 10.1097/01.tp.0000189711.98971.9c. PMID 16421478
- [Background] Kopetz S, Chang GJ, Overman MJ, Eng C, Sargent DJ, Larson DW, Grothey A, Vauthey JN, Nagorney DM, McWilliams RR. Improved survival in metastatic colorectal cancer is associated with adoption of hepatic resection and improved chemotherapy. J Clin Oncol. 2009 Aug 1;27(22):3677-83. doi: 10.1200/JCO.2008.20.5278. Epub 2009 May 26. PMID 19470929
- [Background] Tomlinson JS, Jarnagin WR, DeMatteo RP, Fong Y, Kornprat P, Gonen M, Kemeny N, Brennan MF, Blumgart LH, D'Angelica M. Actual 10-year survival after resection of colorectal liver metastases defines cure. J Clin Oncol. 2007 Oct 10;25(29):4575-80. doi: 10.1200/JCO.2007.11.0833. PMID 17925551
- [Background] Hagness M, Foss A, Line PD, Scholz T, Jorgensen PF, Fosby B, Boberg KM, Mathisen O, Gladhaug IP, Egge TS, Solberg S, Hausken J, Dueland S. Liver transplantation for nonresectable liver metastases from colorectal cancer. Ann Surg. 2013 May;257(5):800-6. doi: 10.1097/SLA.0b013e3182823957. PMID 23360920
- [Background] Dueland S, Hagness M, Line PD, Guren TK, Tveit KM, Foss A. Is Liver Transplantation an Option in Colorectal Cancer Patients with Nonresectable Liver Metastases and Progression on All Lines of Standard Chemotherapy? Ann Surg Oncol. 2015 Jul;22(7):2195-200. doi: 10.1245/s10434-014-4137-0. Epub 2014 Oct 9. PMID 25297902
- [Background] Dueland S, Foss A, Solheim JM, Hagness M, Line PD. Survival following liver transplantation for liver-only colorectal metastases compared with hepatocellular carcinoma. Br J Surg. 2018 May;105(6):736-742. doi: 10.1002/bjs.10769. Epub 2018 Mar 13. PMID 29532908
- [Background] Simoneau E, D'Angelica M, Halazun KJ. Liver transplantation for colorectal liver metastasis. Curr Opin Organ Transplant. 2019 Apr;24(2):175-181. doi: 10.1097/MOT.0000000000000623. PMID 30839338
- [Background] Toso C, Pinto Marques H, Andres A, Castro Sousa F, Adam R, Kalil A, Clavien PA, Furtado E, Barroso E, Bismuth H; Compagnons Hepato-Biliaires Group. Liver transplantation for colorectal liver metastasis: Survival without recurrence can be achieved. Liver Transpl. 2017 Aug;23(8):1073-1076. doi: 10.1002/lt.24791. No abstract available. PMID 28544246
- [Background] Glinka J, Ardiles V, Pekolj J, Mattera J, Sanchez Claria R, de Santibanes E, de Santibanes M. Liver transplantation for non-resectable colorectal liver metastasis: where we are and where we are going. Langenbecks Arch Surg. 2020 May;405(3):255-264. doi: 10.1007/s00423-020-01883-2. Epub 2020 Apr 24. PMID 32333096
- [Background] Dueland S, Grut H, Syversveen T, Hagness M, Line PD. Selection criteria related to long-term survival following liver transplantation for colorectal liver metastasis. Am J Transplant. 2020 Feb;20(2):530-537. doi: 10.1111/ajt.15682. Epub 2019 Nov 28. PMID 31674105